CLINICAL TRIAL: NCT00950937
Title: A Case-control Study to Test the Effects of a Bout of Aerobic Exercise Followed by Resistance Training on Antioxidant System in Human Immunodeficiency Virus (HIV)-Infected and Non-HIV Subjects
Brief Title: Exercise, Oxidative Stress and HIV
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Pedro Dall'Ago, Hospital de Clinicas de Porto Alegre
Other Study IDs: 06067
Record Dates: First submitted 2009-02-16; First posted 2009-08-03 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HIV Group: HIV infected persons
- Control Group: Non HIV-infected persons

SUMMARY:
The purpose of this study is to compare oxidative stress markers and the immunologic characteristics of HIV-infected and non-HIV subjects during a bout of moderate aerobic exercise followed by resistance exercises

ELIGIBILITY:
Inclusion Criteria:

* HIV Group:without contraindications for exercise training; to highly active antiretroviral therapy (HAART) for at least 6 months before enrollment; be classified as low level of physical activity by international physical activity questionnaire (IPAQ) and did not use antioxidant supplements.
* Control Group:negative result for HIV-1 test and the other criteria described above

Exclusion Criteria:

* Subjects with previous history of cardiovascular and neurological disease, diabetes, dyslipidemia, tobacco using, physical disability and pregnant women were excluded from the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants of the HIV group were recruited at the outpatient HIV/AIDS care unit of the Hospital de Clínicas de Porto Alegre (HCPA), whereas the control group (non-HIV) was formed by volunteers of the city of Porto Alegre, Rio Grande do Sul, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2006-06; Primary Completion 2007-01 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Dall'Ago, Professor, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Outpatient HIV/AIDS care unit of the Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV Group | Control Group
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Group | Control Group | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 14 | 14 | 28.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.2 (8.7) | 36 (10.6) | 37.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14.0
  Male | 7 | 7 | 14.0
Region of Enrollment [Number; unit: participants]
  Brazil | 14 | 14 | 28.0

OUTCOME MEASURES:

1. Secondary Outcome: Catalase Activity
Description: Antioxidant activity of the catalase enzyme at three moments: baseline, aerobic and exercise.
Time Frame: 3 times - baseline (before the peak oxygen uptake test), aerobic (immediately after aerobic exercise) and resistance (immediately after resistance exercise).
Measure: Median (Inter-Quartile Range); unit: units of catalase /mg protein
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 14 | 14
units of catalase /mg protein
  Baseline | 0.578 [0.049 to 1.338] | 0.967 [0.312 to 2.322]
  Aerobic | 1.03 [0.316 to 2.598] | 0.855 [0.087 to 1.688]
  Resistance | 0.566 [0.317 to 3.510] | 1.009 [0.333 to 2.096]
Statistical Analysis 1: Comparison: HIV Group vs Control Group; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was utilized to compare the three moments: baseline vs. aerobic, baseline vs. resistance and aerobic vs. resistance
Statistical Analysis 2: Comparison: HIV Group; Test type: Superiority or Other; p < 0.05, Friedman Test; Friedman to compare: baseline vs. aerobic, baseline vs. resistance and aerobic vs. resistance. Wilcoxon was applied to locate the differences
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]

2. Primary Outcome: Total Glutathione
Description: The total glutathione content in erythrocyte concentrate at three moments: baseline, aerobic and resistance exercise.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nmoles glutathione/ ml of sample
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 14 | 14
nmoles glutathione/ ml of sample
  Baseline | 1,964 [319 to 2,577] | 3,490 [597 to 7,596]
  Aerobic | 1,865 [780 to 5,006] | 3,995 [2,308 to 6,068]
  Resistance | 1,767 [516 to 2,420] | 3,206 [2,456 to 7,202]
Statistical Analysis 1: Comparison: HIV Group vs Control Group; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HIV Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Glutathione S-transferase (GST)
Description: Antioxidant activity of the Glutathione S-transferase enzyme at three moments: baseline, aerobic and resistance exercise.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: micromol of GST/min/mg of protein
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 14 | 14
micromol of GST/min/mg of protein
  Baseline | 0.34 [0.18 to 0.58] | 0.5 [0.42 to 0.56]
  Aerobic | 0.34 [0.09 to 0.42] | 0.36 [0.34 to 0.51]
  Resistance | 0.45 [0.31 to 0.63] | 0.46 [0.43 to 0.65]
Statistical Analysis 1: Comparison: HIV Group vs Control Group; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HIV Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]

4. Secondary Outcome: Lipid Peroxidation
Description: Thiobarbituric acid-reactive substances (TBARS) assay was used as an index of lipid peroxidation in erythrocytes, at three moments: baseline, aerobic and resistance exercise.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picomol of TBARS/mg protein
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 14 | 14
picomol of TBARS/mg protein
  Baseline | 2.356 [1.27 to 3.12] | 2.888 [1.118 to 5.002]
  Aerobic | 2.328 [0.909 to 2.922] | 4.164 [2.763 to 6.790]
  Resistance | 2.348 [0.917 to 3.794] | 3.205 [1.753 to 6.840]
Statistical Analysis 1: Comparison: HIV Group vs Control Group; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HIV Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]

5. Secondary Outcome: T CD4
Description: T CD4 lymphocytes counts at three moments: baseline, aerobic and resistance exercise.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Cell/ul of blood
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 14 | 14
Cell/ul of blood
  Baseline | 417 [116 to 1132] | 984 [594 to 2145]
  Aerobic | 428 [70 to 811] | 968 [553 to 1387]
  Resistance | 378 [70 to 981] | 974 [643 to 1411]
Statistical Analysis 1: Comparison: HIV Group vs Control Group; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HIV Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]

6. Secondary Outcome: Neutrophil Count
Description: Neutrophil count at three moments: baseline, aerobic and resistance exercise.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Cell/ul of blood
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 14 | 14
Cell/ul of blood
  Baseline | 3,237 [1,901 to 4,207] | 3,212 [2,328 to 4,174]
  Aerobic | 3,285 [1,610 to 5,476] | 3,476 [2,184 to 9,236]
  Resistance | 3,511 [1,531 to 5,977] | 3,563 [2,422 to 9,214]
Statistical Analysis 1: Comparison: HIV Group vs Control Group; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HIV Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority or Other; p < 0.05, Friedman Test; [statistical method as in outcome 1, analysis 2]

7. Secondary Outcome: Peak Oxygen Uptake
Description: Is the maximum capacity of an individual's body to transport and utilize oxygen during incremental exercise.
Time Frame: 1 time, before the exercise protocol
Measure: Median (Standard Deviation); unit: ml/min
Arm/Group | HIV Group | Control Group
Number analyzed (Participants) | 14 | 14
ml/min | 1,673 (349) | 2,167 (597)
Statistical Analysis 1: Comparison: HIV Group vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Paired t-test was utilized to compare the two groups (HIV group and Control group)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No